CLINICAL TRIAL: NCT05203952
Title: New Therapeutic Approach to Cure Rheumatoid Arthritis
Brief Title: Purify Antigen-specific B Cells From Patients With Rheumatoid Arthritis
Acronym: CURE RA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0735
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Rheumatoid Arthritis
Keywords: B cells; Rheumatoid arthritis; ACPA
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rheumatoid arthritis (RA) is an autoimmune disease characterized by the presence of autoantibodies directed against citrullinated proteins, called ACPAs. These antibodies are very specific to RA, and the severity of the disease is closely correlated with the level of these ACPAs, even though they appear much earlier than the clinical signs. Current treatments by biotherapies are effective but only treat the inflammatory symptoms of the disease or, on the contrary, induce a global immunosuppression with a depletion of all B lymphocytes.

Contrary to the current approaches, the CURE RA project proposes a double innovative character:

* The project aims at specifically destroying B lymphocytes expressing / or secreting ACPAs for a more specific approach to RA, without inducing immunosuppression.
* The new therapeutic molecule is entirely original and has no equivalent at present, it uses the target antigens of autoantibodies, the citrullinated peptides, as tools to destroy the pathogenic B cells that express/produce these autoantibodies.

ELIGIBILITY:
Inclusion criteria:

- Antibodies anti-CCP + (ACPA +) > 250 IU/mL

Exclusion criteria:

* Current or past Rituximab (Mabthera) treatment past (< 9 months)
* Abatacept treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are selected based on the presence of high serum ACPA levels (medical record analyses). Patients treated with Rituximab resulting in total B cell depletion are not selected for this study
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Establishment of B cell line | 1 day
  Establishment of B cell line From first COVID-19 symtpoms, or first positive SARS-COV2 PCR result, to recovery.

SECONDARY OUTCOMES:
Validation of new therapeutic molecules | 1 day
  Validation of new therapeutic molecules

CONTACTS AND LOCATIONS:
Overall Officials: Yves-Marie PERS, MCU-PH, Study Director — University Hospitals of Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC